CLINICAL TRIAL: NCT01144429
Title: Randomized, DB, Parallel Group, MC Study to Evaluate the Efficacy and Safety of Four Doses of Depigmented Glutaraldehyde Polymerized Birch Pollen Allergenic Extract (Depigoid Birch) in Patients With Allergic Rhinitis and/or Rhinoconjunctivitis With or Without Intermittent Asthma
Brief Title: Dose Finding Study for Depigoid Birch: 4 Doses in Patients With Allergic Rhinitis/Rhinoconjunctivitis +-Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leti Pharma GmbH (Industry)
Collaborators: Laboratorios LETI SL (Study Medication) (Unknown); Pierrel Research Europe GmbH (Industry); Labor Dr. Spranger (Central lab) (Unknown)
Responsible Party: Dr. med. Angelika Sager, LETI Pharma GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 603-PG-PSC-173; 2008-008448-26 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Allergic Rhinitis and/or Rhinoconjunctivitis +- Asthma; Immunotherapy, Allergen
Keywords: Allergic Rhinitis +- intermittent asthma; Allergic Rhinoconjunctivitis +- intermittent asthma; Specific Immunotherapy
MeSH Terms: interventions — Allergoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 100 DPP/mL (Active Comparator): Concentration of solution fo s.c. injection: 100 DPP/mL
  Interventions: Biological: Allergoid, allergenic extract of 100% Birch
- 1000 DPP/mL (Active Comparator): Concentration of solution fo s.c. injection: 1000 DPP/mL
  Interventions: Biological: Allergoid, allergenic extract of 100% Birch
- 5000 DPP/mL (Active Comparator): Concentration of solution fo s.c. injection: 5000 DPP/mL
  Interventions: Biological: Allergoid, allergenic extract of 100% Birch
- 10000 DPP/mL (Active Comparator): Concentration of solution fo s.c. injection: 10000 DPP/mL
  Interventions: Biological: Allergoid, allergenic extract of 100% Birch

INTERVENTIONS:
Biological: Allergoid, allergenic extract of 100% Birch — Subcutaneous injections Build-up = 1 day: 0,1mL + 0,2mL + 0,2mL s.c. in intervals on 30 minutes; Maintenance = 5 x single injection of 0,5 mL s.c. every 4 weeks
  Other Names: Depigoid (R); Depigmented, glutaraldehyd-polymerized allergenic extract of

SUMMARY:
Specific immunotherapy for subcutaneous application: Dose finding study to evaluate the correct dose.

4 concentrations of a birch pollen allergen extract are applied in this study. Duration of therapy 20 weeks. Primary criterion is the Conjunctival Provocation Test (CPT), i.e. comparison between treatment arms of increased amount of quantities of allergen to provoke a positive CPT at the end of treatment.

DETAILED DESCRIPTION:
This is a dose finding study and no therapeutic study. Patients will receive in 4-weekly intervals 5x injections of 0,5 ml of a solution of modified birch pollen extract outside the pollen season. The primary endpoint therefore is not the therapeutic effect of the specific immunotherapy (effect on symptoms of allergy during the birch pollen season) but the effect on the CPT. Acc. to the EMEA "Guideline on clinical development of products for specific immunotherapy for the treatment of allergic diseases" provocation tests are accepted as primary outcomes for dose-finding studies.

For the CPT increasing doses of birch pollen solutions are applied to the eye and characteristic symptoms (eye redness, weeping, itching or burning and nose dripping/blockage) are assessed: 0 = absent, 1=mild, 2=moderate, 3=severe). At a score value of >= 5/concentration the test is considered positive and finished.

It is expected that at the end of the study higher doses are necessary to provoke a positive CPT.

Furthermore comparative evaluation of the safety data (AEs) in the different dosage groups is a very important parameter for the evaluation of the outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have provided an appropriately signed and dated informed consent prior to any study specific examination,
2. Patients must be ≥ 18 and ≤ 70 years of age at Visit 1,
3. Patients must have a perception of disease activity of at least 30 mm on a 100 mm visual analogue scale (VAS),
4. Patients must have an FEV1 or PEF value > 80% of the predicted normal value (for PEF: highest result of 3 measurements),
5. Patients must complain about allergic rhinitis and/or rhinoconjunctivitis symptoms for at least 2 years with or without intermittent asthma symptoms, caused by clinical sensitization against birch pollen,
6. IgE-mediated sensitization has to be verified by:

   * suggestive medical history, and
   * specific IgE against birch pollen (CAP-Rast ≥ 2), and
   * a positive SPT to birch pollen (the SPT is considered positive if it results in a wheal diameter of at least 3 mm and at least the size of histamine reference), and
   * a positive CPT with a birch pollen concentration of up to 10,000 SQ-units/mL.

   Special criteria for patients with co-allergies
7. Patients do not suffer from typical symptoms against co-allergens,
8. Specific CAP-RAST against co-allergens < CAP-RAST against birch pollen (the difference has to be ≥ 2), patients with co-allergens against animal dander can be randomized even if the CAP RAST difference is < 2, but must not be exposed to the specific allergen,
9. Result of SPT against co-allergens < result of SPT against birch pollen.

Exclusion Criteria:

1. Acute and chronic conjunctivitis,
2. Infectious conjunctivitis,
3. History of significant clinical manifestations of allergy as a result of sensitization against grass or weed pollen and perennial allergens (e.g. house dust mites),
4. Symptoms due to co-allergies,
5. Persistent asthma, according to the Global Initiative for Asthma (GINA) Guidelines,
6. Acute or chronic inflammatory or infectious airway diseases including recurrent acute or chronic sinusitis,
7. Chronic structural diseases of the lung (e.g. emphysema or bronchiectasis),
8. Diseases of the immune system including autoimmune and immune deficiencies,
9. Any disease, which prohibits the use of adrenaline (e.g. hyperthyroidism),
10. Severe uncontrolled diseases that could increase the risk for the patients participating in the study, which include but are not limited to the following: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases, or hematological disorders,
11. Any malignant disease during the previous 5 years,
12. Any significant abnormal laboratory parameter or alteration in the vital signs that could increase the risk for the study patient,
13. Alcohol, drug, or medication abuse within the past year,
14. Severe psychiatric, psychological, or neurological disorders,
15. Use of immunotherapy against birch pollen within the last 5 years,
16. Topical and systemic treatment with β-blockers,
17. Treatment with substances interfering with the immune system within 1 week prior to Visit 2,
18. Use of tranquillizers or psychoactive drugs within 1 week prior to Visit 1,
19. Use of systemic corticosteroids within 3 months prior to Visit 1,
20. Immunization with vaccines within 7 days prior to Visit 2,
21. Patients with hypersensitivity to excipients of the investigational medicinal product,
22. Patients expected to be non-compliant and/or not co-operative,
23. Exposure to any investigational drug within one month or 6 half lives,
24. Patients who have already participated in this study,
25. Patients who are employees of the institution, or 1st grade relatives, or partners of the investigator,
26. Any donation of germ cells, blood, organs, or bone marrow during the course of the study,
27. Patients who are not contractually capable,
28. Nursing (lactating) women or a positive pregnancy test at Visit 1.
29. Persons who are jurisdictional or governmentally institutionalized.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Conjunctival Provocation Test | At screening and after approx 22 weeks (EoS)
  Comparison between dosage groups of percentage of patients who need an increased amount of allergen to provoke a positive CPT at the end of the treatment (comparison of slope of efficacy) It is expected that at the end of the study higher doses are necessary to provoke a positive CPT.
  Acc. to the EMEA "Guideline on clinical development of products for specific immunotherapy for the treatment of allergic diseases" provocation tests are accepted as primary outcomes for dose-finding studies.

SECONDARY OUTCOMES:
Laboratory parameters (immunology) | At screening and after approx. 22 weeks (EoS)
  specific IgE (Birch), specific IgG1 and IgG4 (Birch). Comparison pre-post will be evaluated
Conjunctival Provocation Test | after approx. 22 weeks
  Analysis of individual results for allergen amount
Laboratory (hematological, clinical chemistry, immunological) as a measure of safety | At screening and after approx. 22 weeks (EoS)
  Clinically relevant changes need to be documented as AE. Comparison pre-post will be displayed descriptively.
Overall assessment of safety (tolerability)at the end of the study | after approx. 22 weeks (EoS)
  At the end of the study investigator and patient will give their general overall impression on the safety of the study treatment on the following scale: excellent (no side effects at all), good (some minor local side effects), moderate (major local side effects or mild systemic side effects) or unaccaptable (anaphylactic reaction).
  Results will be compared between dosage groups
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at 4-weekly intervals (retrospectively at study visits)
  AEs are recorded at the study visits (patients are questioned and the patient diary - where allergy specific symptoms should be recorded by the patients during 48 hrs after each injection of IMP - is assessed by the investigator and AEs recorded in the CRF if applicable) and at any time of the study when site becomes aware of an AE/SAE.
  AE/SAE rate is compared between the treatment groups (safety profile). Also rates of local and systemic reactions will be calculated
Vital signs: Blood pressure and Heart rate as a measure of safety | At screening and every study visit (4-weekly)
  Vital signs are measured a screening and every study visit. Clinically abnormal values must be assessed by the investigator and - if applicable - documented as AE. Vital signs will be evaluated descriptively
Patient diary: Allergy specific symptoms and concomitant medication (rescue m.) for 48 hrs after application of study medication | 48 hrs every 4 weeks after each application of study medication
  Symptoms: urticaria, sneezing, runny nose, cough, dizziness, asthma symptoms, swelling/pain at the injection site.
  Symptoms documented in the diary will be judged and assessed by the investigator and transcribed as AE into the CRF if applicable Medication: Antihistaminics (Eye drops, nose spray), Sultanol, oral corticosteroids, other Intake of medication documented by the patients has to be transcribed to the CRF (Concomitant medication section)
Physical examination acc to local procedures as a measure of safety | At screening and after approx. 22 weeks (EoS)
  A PE has to be performed at screening and end of study visit (22 weeks). Clinically abnormal findings must be assessed by the investigator and documented as AE if applicable. Data will be evaluated descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany; Angelika Sager, Dr., Study Chair — Leti Pharma GmbH, Witten, Germany
Locations (39):
- Germany (25):
  - Dermatology Weber, Augsburg
  - Licca Klinik Dermatologie, Augsburg
  - Allergie-Centrum-Charité, Berlin
  - Klinische Froschung Berlin Mitte, Berlin
  - Hippke, Ear-Nose-Throat Specialist and Allergy, Berlin
  - Universität Bonn, Klinik und Poliklinik für Dermatologie, Bonn
  - Klinikum Carl-Gustav Carus, Klinik+Poliklinik für HNO, Dresden
  - Thieme, Ear-Nose-Throat Specialist and Allergology, Duisburg
  - Dominicus Hautzentrum, Dülmen
  - Spaeth, Ear-Nose-Throat Specialist and Allergy, Düren
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Clinical Research Hamburg GmbH, Hamburg
  - Stefan, Dermatology and Allergy, Hennef (Sieg)
  - Feussner, Pulmology and Allergology, Kassel
  - Tagesklinik für Allergie und Hautkrankheiten Brüning, Kiel
  - Zentrum für Therapiestudien der Innomed Leipzig GmbH, Leipzig
  - Medamed GmbH Studienambulanz, Leipzig
  - Amann, Ear-Nose-Throat Specialist and Allergy, Lingen
  - CRC Universitätsklinikum Mainz, Mainz
  - Universität, Klinik und Poliklinik für Hautkrankheiten, Münster
  - Ear-Nose-Throat Specialist Schaefer, Pirna
  - Palm, Ear-Nose-Throat, Allergology, Röthenbach
  - Steinborn Dermatology, Straubing
  - Zentrum für Rhinologie und Allergie, Wiesbaden
  - Hautarztpraxis Allergie Hoffmann, Witten
- Lithuania (3):
  - Kaunas Distric Hospital, Kaunas
  - Kaunas Medical University Clinics, Kaunas
  - ENT Clinic "Trirema Medica", Vilnius
- Poland (11):
  - Zakład Alergologii, SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Klinika Pulmonologii i Alergologii, SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. N. Barlickiego UM w Łodzi, Lodz
  - NZOZ Centrum Alergologii, Lodz
  - CSK UM w Łodzi, Klinika Immunologii, Reumatologii i Alergii, Zakład Immunologii Klinicznej, Lodz
  - Centrum Alergologii, Poznan
  - Alergologia Plus, Specjalistyczny NZOZ, Ośrodek Diagnostyki i Terapii Uczuleń, Poznan
  - NZOZ Alergo-Med., Poznan
  - Alergo-Med. Specjalistyczna Przychodnia Lekarska Sp. z o. o., Tarnów
  - Poradnia Alergologiczna, Gabinet Lekarski, Tomaszów Mazowiecki
  - NZOZ Almed Specjalistyczna Opieka Medyczna, Wroclaw
  - NZOZ Lekarze Specjaliści J. Małolepszy i Partnerzy, Wroclaw